CLINICAL TRIAL: NCT06375525
Title: Clinical Trial: The Efficacy of Janssen's Icon Application (App) in Improving Adherence to Treatment With Stimulant Medications in Children With Attention Deficit/Hyperactivity Disorder
Acronym: App ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Doron Gothelf MD (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Doron Gothelf MD, Director of Child and Adolescent Psychiatry Unit, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2635-SMC
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Children Aged 6-18 Years With the Diagnosis of ADHD

ARMS (1):
- Application (App), a digital tool (Other): Janssen's icon Application (App), a digital tool designed to improve adherence to medication treatment in children with ADHD.
  Interventions: Device: Janssen's icon Application (App)

INTERVENTIONS:
Device: Janssen's icon Application (App)

SUMMARY:
The overarching aim of the study is to assess the efficacy of Janssen's icon Application (App), a digital tool designed to improve adherence to medication treatment in children with ADHD.

Our specific hypotheses are:

1. In children receiving medication for ADHD those provided with the App tool will be more adherent to treatment than children treated as usual (i.e., not provided with the App tool).
2. Adherent patients will show greater improvement of ADHD symptoms and related dysfunction.

DETAILED DESCRIPTION:
Background and Rationale ADHD is one of the most common neurobehavioral disorders of childhood that affects approximately 6-10% of school-age children and is associated with significant impairment of cognitive and psychosocial functioning (1-3).

Psychostimulant medications are the most effective treatment for ADHD (4). Methylphenidate (MPH) is the drug of choice in Israel for children, adolescents and adults with ADHD and amphetamine derivatives are used when response to MPH is insufficient or when MPH is not tolerable (5).

Without adherence to treatment even the best medication will be ineffective. Adherence is defined as the extent to which a patient's actions correspond to the treatment recommendations of health care providers (6). The literature shows that adherence rates are lower for children as compared to adults, and for psychiatric patients as compared to medical patients (7). As a result, children with psychiatric disorders, such as ADHD, are at great risk for poor medication adherence.

Because of the long-term nature of the treatment, poor adherence turns out to be a crucial issue in ADHD treatment (8). Rates of stimulant adherence in children with ADHD vary considerably across studies but are generally stunningly low. For example, a large community study of urban elementary school children in the Philadelphia area found that only one in five of ADHD children treated with MPH adhered to the treatment (9).

Studies on adherence in children with ADHD suggest that predictors of poor adherence may include older age (10, 11), male gender (12), lower intelligence (12, 13), oppositional-defiant symptoms (13), lower socioeconomic status (14), three-times-daily regimen (10) and the presence of fewer symptoms of ADHD (15). Those who are adherent to their stimulant treatment are more likely to have more severe symptoms (11), high level of knowledge about ADHD, frequent clinical evaluation (16) and lack of proper family support (8).

We believe that the poor adherence to stimulants' treatment in children with ADHD can be improved if we develop intervention programs that focus on increasing adherence to drug treatment. Yet, to the best of our knowledge there are no studies on the efficacy of interventions geared towards improving adherence to medication treatment in children with ADHD.

Objective The overarching aim of the study is to assess the efficacy of Janssen's icon Application (App), a digital tool designed to improve adherence to medication treatment in children with ADHD.

Our specific hypotheses are:

1. In children receiving medication for ADHD those provided with the App tool will be more adherent to treatment than children treated as usual (i.e., not provided with the App tool).
2. Adherent patients will show greater improvement of ADHD symptoms and related dysfunction.

Study Population The study will include 80 children, aged 6-18 years, with the diagnosis of ADHD according to the DSM-5 criteria that are already receiving medication treatment for ADHD with methylphenidate, mixed amphetamine salts, lisdexamfetamine or dexmethylphenidate.

The patients will be consecutively recruited from the Child Psychiatry Unit and ADHD and Learning Disorders Clinic at Edmond & Lili Safra Children's Hospital, Sheba Medical Center.

Inclusion criteria:

1. Diagnosis of ADHD based on the DSM-5;
2. Age between 6 to 18 years
3. Eligible for receiving ADHD treatment with methylphenidate, mixed amphetamine salts, lisdexamfetamine or dexmethylphenidate

3. Parents own smart phone device. 4. Parents will sign a consent form

Study Procedure Diagnostic interviews of children with ADHD and one or both caregivers will be conducted by a child and adolescent psychiatrist. The study will be submitted to the Helsinki committee at the Sheba Medical Center.

The 80 children with ADHD enrolled to this study will be randomized to 2 arms: the study group (n=40) will be provided with the icon App and the control group (n=40) will not be provided the App. The study and control groups will be matched for age, gender distribution, socioeconomic status, and type of ADHD medication. Our plan is to complete the recruitment of subjects within 6 months from study initiation.

The design of the study is also summarized in the Figure and Table below. For all patients an assessment of socio-demographic and clinical characteristics will be conducted at baseline (time 0) by a child and adolescent psychiatrist, using the Attention Module of the Kiddie-SADS (17) and the MINI-KID (18), to screen for symptoms of other comorbid disorders. The ADHD-Rating Scale Questionnaire (ADHD-RS) (19) and the Clinical Global Impression Scale (CGI) (20) will be used to assess the severity of ADHD symptoms and clinical improvement. A research assistant will guide and train the study group families on how to use the App. At the end of months 1, 2 and 3 the patients and their parents will visit the clinic or will be interviewed on the phone, and will be assessed for adherence using the Medication Adherence Rating Scale (MARS) (21) and the Clinician Rating Scale (CRS) (22). In addition, change in ADHD symptoms will be assessed using the ADHD-RS questionnaire, and the CGI. Side effects will be measured using the Barkley Side Effects Rating Scale. Drug accountability will be recorded by the parent as a checkmark on a medication log which will be reviewed by the clinician during the study visits. At the end of visit 3 (after 2 month) we will conduct a Parent Satisfaction Survey.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADHD based on the DSM-5; 2. Age between 6 to 18 years 3. Eligible for receiving ADHD treatment with methylphenidate, mixed amphetamine salts, lisdexamfetamine or dexmethylphenidate 3. Parents own smart phone device. 4. Parents will sign a consent form

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Attention Module of the Kiddie-SADS questionniare | 3 time points: baseline, after 1 month, 3 month after baseline

SECONDARY OUTCOMES:
MINI-KID | 3 time points: baseline, after 1 month, 3 month after baseline

OTHER OUTCOMES:
ADHD-Rating Scale Questionnaire (ADHD-RS) | 3 time points: baseline, after 1 month, 3 month after baseline
Clinical Global Impression Scale (CGI) | 3 time points: baseline, after 1 month, 3 month after baseline
the Barkley Side Effects Rating Scale | 3 time points: baseline, after 1 month, 3 month after baseline
Drug accountability by reviewing the completed medication logs | after 1 month, 3 month after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- ADHD Medical Clinic, Child and Adolescent Psychiatry Unit, Sheba Medical Center, Ramat Gan, Israel